CLINICAL TRIAL: NCT04961125
Title: Multicenter Study on the Pathogenic Germline Gene Variants of Colorectal Polyposis in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-072
Record Dates: First submitted 2021-07-08; First posted 2021-07-14 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Colorectal Polyposis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- colorectal polyposis
  Interventions: Genetic: germline variants

INTERVENTIONS:
Genetic: germline variants — Variants of 139 genes associated with different hereditary cancers and polyposis were screened by next-generation sequencing.

SUMMARY:
Patients suspected of adenomatous polyposis were included. The criteria used were more than 10 polyps observed under colonoscopy, and pathological confirmation of adenoma. Clinical data and pedigree information were collected. The variants of 139 genes associated with different hereditary cancers and polyposis were screened by NGS, which was performed by Genetron Health on the HiSeqX-ten sequencing platform.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of adenomatous polyposis;
2. enough samples (provide at least 5ml of peripheral whole blood) for germline variant detection

Exclusion Criteria:

genetic diagnosis of polyposis syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients suspected of adenomatous polyposis, with more than 10 polyps observed under colonoscopy, and pathological confirmation of adenoma.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-08-02 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
germline variant detection rate in the polyposis population | through study completion, an average of 3 years
  germline variant detection rate in the polyposis population

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - General Hospital of Air Force, Beijing, Beijing Municipality
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - SAHZU, Hangzhou, Zhejinag